CLINICAL TRIAL: NCT05784077
Title: Prevalenza Delle Apnee Notturne e Riduzione Dei Fattori Promotori Nella Fibrillazione Atriale
Brief Title: PRevalence of Obstructive Sleep apnoEa and Reduction of Promoters in AF
Acronym: PROSERPin-AF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09C020
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation; Osa Syndrome
MeSH Terms: conditions — Atrial Fibrillation; Carnevale syndrome | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Polysomnography — Study of the sleep pattern
Behavioral: Lifestyle counselling — Weight loss counselling

SUMMARY:
This study aims to identify how many patients who have atrial fibrillation, also have sleep apnoea. This is important because sleep apnoea can be a trigger to atrial fibrillation and it can be corrected with a simple intervention. Therefore it is important to understand its prevalence (how many patients with atrial fibrillation are affected by it). Also, obesity and sleep disorders are often associated, therefore the evolution of atrial fibrillation is studied in patients who also have obesity and have lost weight compared with patients who did not loose any weight or are not obese. As medications or therapy are not changed, this is an observational study.

ELIGIBILITY:
Inclusion Criteria primary outcome:

* 1 episode of atrial fibrillation in the previous year

Inclusion Criteria secondary outcome:

* BMI > o = 27Kg/m2
* AHI >30 o con 15<AHI<30 associated with other symptoms (sleeplessness, uncontrolled hypertension and cerebral events)

Exclusion Criteria:

* Ejection Fraction <50%
* HFpEF not related to atrial fibrillation.
* coronary artery disease
* valvular cardiomyopathy
* patient already in treatment for sleep apnoea
* hyperthyroidism

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients between 18 and 75 years of age, male and female, who come to the study centre between January 2019 and January 2023 with a diagnosis of atrial fibrillation and a recurrence (or first episode) in the previous year and who can undergo polysomnography
Sampling Method: Probability Sample
Enrollment: 343 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in prevalence of obstructive sleep apnoea in patients with atrial fibrillation | Baseline and at 3, 6, 12, 24 and 36 months
  Change in prevalence of obstructive sleep apnoea from baseline to 3 years
Percentage of men and women with obstructive sleep apnoea in patients with atrial fibrillation | Baseline
  Percentage of men and women with obstructive sleep apnoea in patients with atrial fibrillation

SECONDARY OUTCOMES:
Change in body weight | Baseline and at 3, 6, 12, 24 and 36 months
  Change in body weight from baseline to 3 years
Change in incidence of atrial fibrillation recurrencies | Baseline and at 3, 6, 12, 24 and 36 months
  Change in incidence of atrial fibrillation recurrencies from baseline to 3 years
Change in quality of life | Baseline and at 3, 6, 12, 24 and 36 months
  Change in quality of life from baseline to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy